CLINICAL TRIAL: NCT01999868
Title: Efficacy of Ustekinumab (Anti-IL-12/23) Followed by Abatacept (CTLA4-Ig) for the Treatment of Psoriasis Vulgaris (ITN059AI)
Brief Title: Efficacy of Ustekinumab Followed by Abatacept for the Treatment of Psoriasis Vulgaris
Acronym: PAUSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ITN059AI
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: psoriasis vulgaris; ustekinumab; abatacept
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab; Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UST, ABA/UST Placebo (Experimental): Participants received 2 subcutaneous injections of open-label ustekinumab (UST) (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and were then randomized to receive blinded (masked) treatment of abatacept (ABA) (125 mg) subcutaneous injections weekly from Week 12 to 39, in addition to ustekinumab placebo subcutaneous injections at Weeks 16 and 28.
  Interventions: Biological: Ustekinumab; Biological: Abatacept; Drug: UST Placebo
- UST, UST/ABA Placebo (Active Comparator): Participants received 2 subcutaneous injections of open-label ustekinumab (UST) (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and were then randomized to receive blinded (masked) treatment of ustekinumab (45 mg if <=100 kg or 90 mg if >100 kg at study entry) subcutaneous injections at Weeks 16 and 28, in addition to abatacept (ABA) placebo subcutaneous injections weekly from Week 12 to 39.
  Interventions: Biological: Ustekinumab; Drug: ABA Placebo

INTERVENTIONS:
Biological: Ustekinumab — Ustekinumab interferes with the actions of proteins, interleukin 12 (IL12) and interleukin 23 (IL23), which reduces inflammation (swelling) in the skin. Stelara™ is the trade name for ustekinumab and is approved by the U.S. Food and Drug Administration (FDA) to treat psoriasis.
  Dose:
  Participants who weigh <= 100 kg at study entry will receive 45 mg of ustekinumab.
  Participants who weigh > 100 kg at study entry will receive 90 mg of ustekinumab.
  Other Names: anti-IL-12/23; Stelara
Biological: Abatacept — Abatacept (one form of the protein called CTLA4-Ig) interacts with the immune system, reducing the activity of T-cells and may prevent relapse. Orencia™ is the trade name for abatacept, and it is approved by the FDA to treat rheumatoid arthritis in adults.
  Dose:
  125 mg sub-cutaneous injection
  Other Names: CTLA4-Ig; cytotoxic T lymphocyte antigen immunoglobulin fusion protein; Orencia
  Arms: UST, ABA/UST Placebo
Drug: UST Placebo — The abatacept treatment group will also receive subcutaneous placebo for ustekinumab (sterile normal saline) at week 16 and week 28, corresponding to the ustekinumab dosing regimen.
  Other Names: Placebo for Ustekinumab; Ustekinumab Placebo
  Arms: UST, ABA/UST Placebo
Drug: ABA Placebo — The ustekinumab treatment group will also receive weekly subcutaneous injections of placebo for abatacept from week 12 to week 39, corresponding to the abatacept dosing regimen.
  Other Names: Placebo for Abatacept; Abatacept Placebo
  Arms: UST, UST/ABA Placebo

SUMMARY:
The purpose of this study is to determine if the use of ustekinumab, followed by abatacept, will prevent relapse in people with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic immune disease of the skin and joints that affects about 2% of the population. The most common form of psoriasis is plaque psoriasis, also called psoriasis vulgaris. A variety of drugs, including biologics, are available for treatment of moderate to severe psoriasis. When biologic agents are stopped, psoriasis can return (relapse) and often requires the biologic to be restarted and continued. No treatment program has been identified to prevent relapse of psoriasis.

The study design has a lead-in period of weight-based ustekinumab treatment, with all participants receiving either 45 mg ustekinumab (<= 100 kg) or 90 mg ustekinumab (> 100 kg) administered subcutaneously at weeks 0 and 4. At week 12, participants will be assessed for a Psoriasis Area and Severity Index (PASI) 75 response to ustekinumab. Participants who do not achieve a PASI 75 score will be discontinued from the investigation and permitted to seek standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of plaque psoriasis for at least 6 months
* Baseline Psoriasis Area and Severity Index (PASI) score >= 12
* >=10% body surface area psoriasis involvement
* Willingness to forgo other available psoriasis therapies, live vaccines, and pregnancy during the trial
* Ability and willingness to provide informed consent and comply with study requirements

Exclusion Criteria:

* Non-plaque forms of psoriasis
* Grade 2 or 3 moderate to severe psoriatic arthritis not adequately managed with non-steroidal anti-inflammatory drugs (NSAIDs)
* Myocardial infarction, unstable angina, cerebrovascular accident, or other significant cardiovascular event within the previous one year
* Chronic obstructive pulmonary disease (COPD)
* Comorbid condition that requires regular systemic corticosteroid treatment
* History of malignancy, except treated basal cell skin carcinoma
* Treated basal cell skin carcinoma within the previous 5 years
* Severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease, or any other medical condition that, in the investigator's opinion, places the participant at risk by participating in this study
* History of recent or ongoing uncontrolled bacterial, viral, fungal, or other opportunistic infections
* Evidence of infection with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV)
* Positive QuantiFERON-TB Gold test. Purified Protein Derivative (PPD) tuberculin test may be substituted for QuantiFERON-TB Gold test.
* Severe reaction or anaphylaxis to any human monoclonal antibody
* Any previous treatment with agents targeting Interleukin (IL)-12 or IL-23, including ustekinumab
* Any previous treatment with abatacept
* Treatment with biologic agents within previous 3 months, including adalimumab, etanercept, and infliximab
* Treatment with immunosuppressive medications, including methotrexate, cyclosporine, oral retinoids, prednisone, or phototherapy within previous 4 weeks
* Topical psoriasis treatment within previous 2 weeks, including topical corticosteroids, vitamin D analogues, retinoids, calcineurin inhibitors, salicylic acid, and coal tar
* Investigational study medication within previous 6 months
* Liver function test (aspartate aminotransferase [AST], alanine aminotransferase [ALT], or alkaline phosphatase) results that are >/= 2x the upper limit of normal (ULN).
* Serum creatinine >= 2x the ULN.
* Any of the following hematologic abnormalities, confirmed by repeat test at least 1 week apart:

  1. White blood count <3,000/μL or >14,000/μL;
  2. Lymphocyte count <1,000/μL;
  3. Neutrophil count <1,500/μL;
  4. Platelet count <150,000 /μL; or
  5. Hemoglobin <10 g/dL.
* Females who are pregnant, lactating, planning on pregnancy during the study period, or unwilling to use FDA-approved method of birth control
* Receipt of a live vaccine (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, and smallpox) in the 6 weeks before enrollment
* BCG (Bacillus Calmette-Guérin) vaccine one year prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, PhD, Principal Investigator — The Rockefeller University
Locations (10):
- United States (8):
  - Dermatology Research Associates, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Tulane University School of Medicine: Dept. of Dermatology, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - The Rockefeller University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western University, Cleveland, Ohio
  - The University of Utah, Salt Lake City, Utah
- Canada (2):
  - Kirk Barber Research, Calgary, Alberta
  - Innovaderm Research Inc., Montreal, Quebec

REFERENCES:
- [Derived] Harris KM, Smilek DE, Byron M, Lim N, Barry WT, McNamara J, Garcet S, Konrad RJ, Stengelin M, Bathala P, Korman NJ, Feldman SR, Boh EE, Barber K, Laumann AE, Helfrich YR, Krueger GG, Sofen H, Bissonnette R, Krueger JG. Effect of Costimulatory Blockade With Abatacept After Ustekinumab Withdrawal in Patients With Moderate to Severe Plaque Psoriasis: The PAUSE Randomized Clinical Trial. JAMA Dermatol. 2021 Nov 1;157(11):1306-1315. doi: 10.1001/jamadermatol.2021.3492. PMID 34643650
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- See also: PAUSE (ITN059AI) ITN Study website — http://www.pausestudy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 148 participants were screened and 108 of those participants were enrolled at 8 sites in the US and 2 sites in Canada between March 2014 and April 2016
Pre-assignment Details: Enrolled participants received open-label ustekinumab in the lead-in phase (Week 0 to 12). Participants with at least 75% reduction in Psoriasis Area Severity Index (PASI) score at Week 12 compared to Week 0 were eligible for the blinded treatment phase (Week 12 to 40).
Groups:
- Ustekinumab, Abatacept + Ustekinumab Placebo: Participants received 2 subcutaneous injections of open-label ustekinumab (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and received blinded treatment of abatacept (125 mg) subcutaneous injections weekly from Week 12 to 39, in addition to ustekinumab placebo subcutaneous injections at Weeks 16 and 28.
- Ustekinumab, Ustekinumab + Abatacept Placebo: Participants received 2 subcutaneous injections of open-label ustekinumab (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and received blinded treatment of ustekinumab (45 mg if <=100 kg or 90 mg if >100 kg at study entry) subcutaneous injections at Weeks 16 and 28, in addition to abatacept placebo subcutaneous injections weekly from Week 12 to 39.
- Ustekinumab, Not Randomized: Participants received 2 subcutaneous injections of open-label ustekinumab (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase but were not randomized to a blinded treatment group.
Period: Lead-in Phase (Week 0 - 12)
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo | Ustekinumab, Not Randomized
Started | 45 | 46 | 17
Completed | 45 | 46 | 12
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 5
Period: Blinded Treatment Phase (Week 12 - 40)
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo | Ustekinumab, Not Randomized
Started | 45 | 46 | 0 (Participants didn't meet eligibility requirements for randomization or withdrew prior to Week 12.)
Completed | 27 | 35 | 0
Not Completed | 18 | 11 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Met study drug Discontinuation Criteria | 1 | 2 | 0
Not completed — Met psoriasis relapse criterion | 8 | 1 | 0
Not completed — Transportation issues | 1 | 0 | 0
Not completed — Worsening psoriasis | 4 | 0 | 0
Period: Blinded Observation Phase (Week 40 - 88)
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo | Ustekinumab, Not Randomized
Started | 27 | 35 | 0
Completed | 4 | 6 | 0
Not Completed | 23 | 29 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Met psoriasis relapse criterion | 10 | 19 | 0
Not completed — Terminated early from study in error | 0 | 2 | 0
Not completed — Worsening psoriasis | 12 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Subjects that signed informed consent, were eligible for the study, and were administered at least one dose of open-label ustekinumab in the lead-in phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo | Ustekinumab, Not Randomized | Total
Number analyzed (Participants) | 45 | 46 | 17 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (10.5) | 44.1 (11.8) | 42.8 (15.0) | 46.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 3 | 35
  Male | 27 | 32 | 14 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 2 | 12
  Not Hispanic or Latino | 42 | 39 | 15 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 0 | 6
  White | 36 | 42 | 17 | 95
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 14 | 6 | 35
  United States | 30 | 32 | 11 | 73
Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Psoriasis Area Severity Index (PASI) score was the score assessed at Week 0. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
  units on a scale | 19.2 (8.1) | 20.0 (8.2) | 21.2 (7.7) | 19.9 (8.1)
Psoriasis Area Severity Index (PASI) (Randomization Strata) [Count of Participants; unit: Participants] — Number of participants with low and high Psoriasis Area Severity Index (PASI) scores. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). Scores of 12-20 were considered "low" and scores >20, "high."
  Participants
    Low (12 - 20) | 31 | 32 | 8 | 71
    High (>20) | 14 | 14 | 9 | 37
Physician's Global Assessment (PGA) Score [Mean (Standard Deviation); unit: units on a scale] — The Physician's Global Assessment (PGA) is an overall assessment of psoriasis severity. Duration, erythema and scaling are assessed, averaged, and given a score ranging from 0 to 5 based on the majority of the psoriatic lesions, with higher scores indicating worse disease. A PGA average score < 1.5 was classified as "cleared or minimal."
  units on a scale | 3.5 (0.7) | 3.3 (0.5) | 3.5 (0.6) | 3.4 (0.6)
Physician's Global Assessment (PGA) Score (Categorical) [Count of Participants; unit: Participants] — Number of participants with "cleared or minimal" average Physician's Global Assessment (PGA) scores and those with average PGA scores worse than minimal. The Physician's Global Assessment (PGA) is an overall assessment of psoriasis severity. Duration, erythema and scaling are assessed, averaged, and given a score ranging from 0 to 5 based on the majority of the psoriatic lesions, with higher scores indicating worse disease. A PGA average score < 1.5 was classified as "cleared or minimal."
  Participants
    Cleared or Minimal (PGA <1.5) | 0 | 0 | 0 | 0
    Worse than Minimal (PGA ≥ 1.5) | 45 | 46 | 17 | 108
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — Dermatology Life Quality Index (DLQI) is a 10-question, participant-reported questionnaire assessing quality of life with respect to skin conditions in the areas of Symptoms and Feelings; Daily Activities; Leisure; Work and School; Personal Relationships; and Treatment. Each question measures the effect the skin condition has on a participant's quality of life. Responses range from "Not at all" (score = 0) to "Very much" (score = 3). The overall score is the sum for all 10 questions and ranges from 0-30, with higher scores indicating a poor quality of life.
  units on a scale | 14.2 (8.1) | 13.5 (7.0) | 13.5 (8.8) | 13.8 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Psoriasis Relapse (Treating Drop-Outs as Relapse)
Description: The percentage of participants who experienced psoriasis relapse in the interval from Week 12 to 88. Psoriasis relapse is defined as loss of ≥ 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at Week 12. This occurs if the participant obtains a PASI score at any evaluation during the specified time interval that is ≥ Week 12 PASI + [(Baseline PASI -Week 12 PASI)/2]). Participants who terminated early from the study (drop-outs) were considered to have experienced relapse at time of drop-out. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
Time Frame: Post-randomization (Week 12 to 88)
Population: The intent-to-treat population includes all participants who were found to be eligible after the 12-week lead-in period and underwent random assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
percentage of participants
  Week 12-88 | 91.1 | 87.0
  Week 12-40 | 55.6 | 30.4
  Week 28-88: number analyzed (Participants) | 36 | 38
  Week 28-88 | 88.9 | 84.2
  Week 40-88: number analyzed (Participants) | 26 | 36
  Week 40-88 | 84.6 | 83.3
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88. This interval corresponds to the time from randomization until the end of the study. This analysis is the primary analysis of the primary endpoint; Test type: Superiority; p = 0.41, Regression, Logistic — Two-sided test; Randomization stratum (PASI score at week 0: 12-20 or >20) and duration of disease prior to screening, centered about the median, are covariates
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40. This interval corresponds to the time from randomization until the end of the blinded treatment phase; Test type: Superiority; p = 0.013, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 28 to 88. This interval corresponds to the time from the last scheduled dose of ustekinumab or ustekinumab placebo until the end of the study; Test type: Superiority; p = 0.50, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 40 to 88. This interval corresponds to the time from the beginning of the blinded observation phase until the end of the study; Test type: Superiority; p = 0.67, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Who Experienced Psoriasis Relapse (Treating Drop-Outs as No Relapse)
Description: The percentage of participants who experienced psoriasis relapse in the interval from Week 12 to 88. Psoriasis relapse is defined as loss of ≥ 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at Week 12 (Baseline PASI -Week 12 PASI). Participants who terminated early from the study due to reasons other than psoriasis relapse or worsening psoriasis (drop-outs) were considered to have not experienced relapse at time of drop-out. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
Time Frame: Post-randomization (Week 12 to 88)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
percentage of participants
  Week 12-88 | 75.6 | 52.2
  Week 12-40 | 42.2 | 10.9
  Week 28-88: number analyzed (Participants) | 36 | 38
  Week 28-88 | 83.3 | 60.5
  Week 40-88: number analyzed (Participants) | 26 | 36
  Week 40-88 | 80.8 | 63.9
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88. This interval corresponds to the time from randomization until the end of the study; Test type: Superiority; p = 0.019, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40. This interval corresponds to the time from randomization until the end of the blinded treatment phase; Test type: Superiority; p = 0.001, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.018, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.07, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Experienced Psoriasis Relapse (Treating Drop-Outs as Missing Relapse Status)
Description: The percentage of participants who experienced psoriasis relapse in the interval from Week 12 to 88. Psoriasis relapse is defined as loss of ≥ 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at Week 12 (Baseline PASI -Week 12 PASI). Participants who terminated early due to reasons other than psoriasis relapse or worsening psoriasis were considered to have a missing relapse status at time of drop-out and were excluded from the analyses. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
Time Frame: Post-randomization (Week 12 to 88)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
percentage of participants
  Week 12-88: number analyzed (Participants) | 38 | 30
  Week 12-88 | 89.5 | 80.0
  Week 12-40: number analyzed (Participants) | 39 | 37
  Week 12-40 | 48.7 | 13.5
  Week 28-88: number analyzed (Participants) | 34 | 29
  Week 28-88 | 88.2 | 79.3
  Week 40-88: number analyzed (Participants) | 25 | 29
  Week 40-88 | 84.0 | 79.3
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88. This interval corresponds to the time from randomization until the end of the study; Test type: Superiority; p = 0.16, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40. This interval corresponds to the time from randomization until the end of the blinded treatment phase; Test type: Superiority; p = 0.002, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.23, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.43, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Psoriasis Relapse (Treating Drop-Outs as Relapse)
Description: Time in weeks from Week 12 to psoriasis relapse. Psoriasis relapse is defined as loss of ≥ 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at Week 12. This occurs if the participant obtains a PASI score at any evaluation during the specified time interval that is ≥ Week 12 PASI + [(Baseline PASI -Week 12 PASI)/2]). Participants who terminated early from the study (drop-outs) were considered to have experienced relapse at time of drop-out. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
Time Frame: Post-randomization (Week 12 to 88)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
weeks | 28 [24 to 40] | 40 [32 to 44]
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88. This interval corresponds to the time from randomization until the end of the study; Test type: Superiority; p = 0.06, Grouped survival analysis — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40. This interval corresponds to the time from randomization until the end of the blinded treatment phase; Test type: Superiority; p = 0.008, Grouped survival analysis — Two-sided test; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Psoriasis Relapse (Treating Drop-Outs as Censored)
Description: Time in weeks from Week 12 to psoriasis relapse. Psoriasis relapse is defined as loss of ≥ 50% of the initial Psoriasis Area and Severity Index (PASI) improvement measured at Week 12. This occurs if the participant obtains a PASI score at any evaluation during the specified time interval that is ≥ Week 12 PASI + [(Baseline PASI -Week 12 PASI)/2]). Participants who terminated early from the study due to reasons other than psoriasis relapse or worsening psoriasis (drop-outs) were censored at the time of drop-out. PASI is an assessment for psoriasis severity based on 4 body areas: Head and Neck, Upper Extremities, Trunk, and Lower Extremities. Psoriasis severity within each body area is assessed for Redness (score 0-4), Thickness (score 0-4) and Scaling (score 0-4). Scores for each body area are summed and weighted by the affected Body Surface Area (score 0-6) to produce the total score. The score ranges from 0 (no psoriasis present) to 72 (very severe psoriasis).
Time Frame: Post-randomization (Week 12 to 88)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
weeks | 28 [28 to 40] | 48 [44 to 56]
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88. This interval corresponds to the time from randomization until the end of the study; Test type: Superiority; p = 0.005, Grouped survival analysis — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40. This interval corresponds to the time from randomization until the end of the blinded treatment phase; Test type: Superiority; p = 0.001, Grouped survival analysis — Two-sided test; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Were Cleared or Minimal in the Physician's Global Assessment (PGA)
Description: Percentage of participants who were classified as cleared or minimal in the Physician's Global Assessment (PGA) average score at the specified post-randomization time point. The PGA assesses the severity of the psoriasis in 3 components: induration, erythema and scaling. Each component is given a score ranging from 0 to 5 based on the majority of the participant's psoriasis lesions, with higher scores indicating worse disease. A PGA average score < 1.5 was classified as "cleared or minimal."
Time Frame: Week 40, Week 88
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
percentage of participants
  Week 40: number analyzed (Participants) | 26 | 34
  Week 40 | 26.9 | 58.8
  Week 88: number analyzed (Participants) | 4 | 6
  Week 88 | 75.0 | 50.0
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 40; Test type: Superiority; p = 0.013, Regression, Logistic — Two-sided test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 88; Test type: Superiority; p = 0.95, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI)
Description: Change in the Dermatology Life Quality Index (DLQI) score from Week 12 to the specified post-randomization time point. DLQI is a 10-question, participant-reported questionnaire that assesses quality of life with respect to skin conditions in the areas of symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Each question measures the level of effect that the skin condition has on quality of life, and responses range from 'Not at all' (score = 0) to 'Very much' (score = 3). The overall score is the sum of the scores for all 10 questions and ranges from 0-30, with higher scores indicating worse quality of life.
Time Frame: Week 40, Week 88
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
Units on a Scale
  Week 40: number analyzed (Participants) | 26 | 34
  Week 40 | 2.2 (5.3) | 0.6 (3.9)
  Week 88: number analyzed (Participants) | 4 | 6
  Week 88 | -4.3 (3.7) | 0.0 (2.1)
Statistical Analysis 1: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 40; Test type: Superiority; p = 0.18, ANCOVA — Two-sided test; Randomization stratum (PASI score at week 0: 12-20 or >20), baseline DLQI, and pre-screening disease duration, centered on the median, are covariates
Statistical Analysis 2: Comparison: Ustekinumab, Abatacept + Ustekinumab Placebo vs Ustekinumab, Ustekinumab + Abatacept Placebo; Week 12 to 88; Test type: Superiority; p = 0.045, ANCOVA — Two-sided test; Randomization (PASI score week 0:12-20 or >20), DLQI score at baseline, duration of disease prior to screening, centered about median, are covariates

8. Secondary Outcome: Frequency and Severity of Adverse Events and Serious Adverse Events (By Participant, Lead-in Phase)
Description: Number of participants who experienced adverse events (AEs) during the lead-in phase (Week 0 to 12), classified by severity and type. AEs were classified by grade according to the National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03, and all Grade 2 or greater AEs were collected in the database. In addition, new onset or worsening psoriatic arthritis was separately collected and graded from 1 to 3 along a study-specific functional scale. AEs were also classified based on relatedness to study drug, whether they led to study drug discontinuation, and whether they were AEs of special interest as specified in the protocol.
Time Frame: Lead-In Phase (Week 0 to 12)
Population: The safety population includes all participants who received at least one dose of treatment after enrollment.
Measure: Number; unit: Number of participants
Groups:
- Safety: The safety population includes all participants who received at least one dose of treatment after enrollment.
Arm/Group | Safety
Number analyzed (Participants) | 108
Number of participants
  All AEs | 30
  AEs indicated as serious | 2
  AEs with an outcome of death | 0
  AEs of special interest | 0
  Grade 2 AEs | 28
  Grade 3 AEs | 2
  Grade 4 AEs | 0
  Grade 1 Psoriatic Arthritis AEs | 2
  Grade 2 Psoriatic Arthritis AEs | 0
  Grade 3 Psoriatic Arthritis AEs | 0
  AEs that lead to study drug discontinuation | 0
  AEs related to open label Ustekinumab | 11

9. Secondary Outcome: Frequency and Severity of Adverse Events and Serious Adverse Events (By Event, Lead-in Phase)
Description: Number of adverse events (AEs) that occurred during the lead-in phase (Week 0 to 12), classified by severity and type. AEs were classified by grade according to the National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03, and all Grade 2 or greater AEs were collected in the database. In addition, new onset or worsening psoriatic arthritis was separately collected and graded from 1 to 3 along a study-specific functional scale. AEs were also classified based on relatedness to study drug, whether they led to study drug discontinuation, and whether they were AEs of special interest as specified in the protocol.
Time Frame: Lead-In Phase (Week 0 to 12)
Population: The safety population includes all participants who received at least one dose of treatment after enrollment.
Measure: Number; unit: Number of Events
Arm/Group | Safety
Number analyzed (Participants) | 108
Number of Events
  All AEs | 51
  AEs indicated as serious | 2
  AEs with an outcome of death | 0
  AEs of special interest | 0
  Grade 2 AEs | 47
  Grade 3 AEs | 2
  Grade 4 AEs | 0
  Grade 1 Psoriatic Arthritis AEs | 2
  Grade 2 Psoriatic Arthritis AEs | 0
  Grade 3 Psoriatic Arthritis AEs | 0
  AEs that lead to study drug discontinuation | 0
  AEs related to open label Ustekinumab | 20

10. Secondary Outcome: Frequency and Severity of Adverse Events and Serious Adverse Events (By Participant, Post-Randomization)
Description: Number of participants who experienced adverse events (AEs) during the post-randomization phase (Week 12 to 100), classified by severity and type. AEs were classified by grade according to the National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03, and all Grade 2 or greater AEs were collected in the database. In addition, new onset or worsening psoriatic arthritis was separately collected and graded from 1 to 3 along a study-specific functional scale. AEs were also classified based on relatedness to study drug, whether they led to study drug discontinuation, and whether they were AEs of special interest as specified in the protocol. AEs that started prior to randomization but became serious after randomization were included in the counts for the post-randomization time period.
Time Frame: From randomization (Week 12) to last safety follow-up visit (up to Week 100)
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
Number of participants
  All AEs | 28 | 22
  AEs indicated as serious | 2 | 5
  AEs with an outcome of death | 0 | 0
  AEs of special interest | 2 | 1
  Grade 2 AEs (CTCAE) | 27 | 20
  Grade 3 AEs (CTCAE) | 4 | 7
  Grade 4 AEs (CTCAE) | 0 | 2
  Grade 1 Psoriatic Arthritis AEs | 0 | 0
  Grade 2 Psoriatic Arthritis AEs | 2 | 1
  Grade 3 Psoriatic Arthritis AEs | 0 | 0
  AEs that lead to study drug discontinuation | 1 | 2
  AEs related to open-label Ustekinumab | 5 | 8
  AEs related to Ustekinumab/Ustekinumab Placebo | 7 | 9
  AEs related to Abatacept/Abatacept Placebo | 11 | 11

11. Secondary Outcome: Frequency and Severity of Adverse Events and Serious Adverse Events (By Event, Post-Randomization)
Description: Number of adverse events (AEs) that occurred during the post-randomization phase (Week 12 to 100), classified by severity and type. AEs were classified by grade according to the National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03, and all Grade 2 or greater AEs were collected in the database. In addition, new onset or worsening psoriatic arthritis was separately collected and graded from 1 to 3 along a study-specific functional scale. AEs were also classified based on relatedness to study drug, whether they led to study drug discontinuation, and whether they were AEs of special interest as specified in the protocol. AEs that started prior to randomization but became serious after randomization were included in the counts for the post-randomization time period.
Time Frame: From randomization (Week 12) to last safety follow-up visit (up to Week 100)
Population: as for outcome 1
Measure: Number; unit: Number of Events
Arm/Group | Ustekinumab, Abatacept + Ustekinumab Placebo | Ustekinumab, Ustekinumab + Abatacept Placebo
Number analyzed (Participants) | 45 | 46
Number of Events
  All AEs | 59 | 59
  AEs indicated as serious | 2 | 9
  AEs with an outcome of death | 0 | 0
  AEs of special interest | 2 | 1
  Grade 2 AEs (CTCAE) | 53 | 47
  Grade 3 AEs (CTCAE) | 4 | 7
  Grade 4 AEs (CTCAE) | 0 | 4
  Grade 1 Psoriatic Arthritis AEs | 0 | 0
  Grade 2 Psoriatic Arthritis AEs | 2 | 1
  Grade 3 Psoriatic Arthritis AEs | 0 | 0
  AEs that lead to study drug discontinuation | 1 | 3
  AEs related to open-label Ustekinumab | 5 | 11
  AEs related to Ustekinumab/Ustekinumab Placebo | 9 | 17
  AEs related to Abatacept/Abatacept Placebo | 15 | 20

ADVERSE EVENTS:
Time Frame: Week 0 to Week 100
Groups:
- UST Open Label: Participants received 2 subcutaneous injections of open-label ustekinumab (UST) (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase.
- Post Randomization: UST, ABA/UST Placebo: Participants received 2 subcutaneous injections of open-label ustekinumab (UST) (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and received blinded treatment of abatacept (ABA) (125 mg) subcutaneous injections weekly from Week 12 to 39, in addition to ustekinumab placebo subcutaneous injections at Weeks 16 and 28.
- Post Randomization: UST, UST/ABA Placebo: Participants received 2 subcutaneous injections of open-label ustekinumab (UST) (45 mg for participants weighing <=100 kg at study entry or 90 mg for those weighing >100 kg at study entry), at Weeks 0 and 4 during the lead-in phase and received blinded treatment of ustekinumab (45 mg if <=100 kg or 90 mg if >100 kg at study entry) subcutaneous injections at Weeks 16 and 28, in addition to abatacept (ABA) placebo subcutaneous injections weekly from Week 12 to 39.
Arm/Group | UST Open Label | Post Randomization: UST, ABA/UST Placebo | Post Randomization: UST, UST/ABA Placebo
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/108 | 2/45 | 5/46
Other Adverse Events (participants affected / at risk) | 4/108 | 6/45 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UST Open Label (N=108) | Post Randomization: UST, ABA/UST Placebo (N=45) | Post Randomization: UST, UST/ABA Placebo (N=46)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UST Open Label (N=108) | Post Randomization: UST, ABA/UST Placebo (N=45) | Post Randomization: UST, UST/ABA Placebo (N=46)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT01999868/Prot_SAP_000.pdf